CLINICAL TRIAL: NCT05804539
Title: The Recovering Strategy on Forward Head Posture in Chinese Adolescents With Explainable Artificial Intelligence: Tai Chi and Manual Therapy
Brief Title: The Recovering Strategy on Forward Head Posture in Chinese Adolescents: Tai Chi and Manual Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Normal University (Other)
Responsible Party: Principal Investigator, Guang Yang, Prof. Dr., Prof.Dr., Northeast Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CCEE2021
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Forward Head Posture
Keywords: forward head posture
MeSH Terms: interventions — Musculoskeletal Manipulations; Tai Ji

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual therapy (Experimental): Each lesson has a duration of 40 minutes, including the first five minutes of warm-up, 30 minutes of manual therapy and the last five minutes of cool-down.
  Interventions: Behavioral: Manual therapy
- Tai Chi (Experimental): Each lesson has a duration of 40 minutes, including the first five minutes of warm-up, 30 minutes of Tai Chi and the last five minutes of cool-down.
  Interventions: Behavioral: Tai Chi
- Tai Chi and Manual therapy (Experimental): Each lesson has a duration of 40 minutes, including the first five minutes of warm-up, 15-min Tai Chi exercise and 15-min manual therapy, with the order of intervention being Tai Chi exercise first and then manual therapy, and the last five minutes of cool-down.
  Interventions: Behavioral: Tai Chi and Manual therapy

INTERVENTIONS:
Behavioral: Manual therapy — The therapist checks the range of motion of the cervical joints and gives manual treatment to the restricted joints. Throughout the examination, the subject lied in a supine position on a professional rehabilitation bed with the seventh cervical vertebra (C7) on the edge of the bed and the other the body above the C7 were placed off the bed. The therapist held the subject's occipital bone with one hand and the radial aspect of the second metacarpophalangeal joint of the other hand to grip the spinous process of the sixth cervical vertebra and slowly pushed the occiput downward to check the joint mobility of the fifth cervical vertebra and the sixth cervical vertebra. After the examination, the restricted joint was accurately located and treated with targeted manual therapy. For example, stretching was performed with the right side of C4-C5 flexed, closing only the right side of the subject's C4-C5 as much as possible to increase joint mobility on the right side of C4-C5.
  Arms: Manual therapy
Behavioral: Tai Chi — Based on the characteristics of young people and the need to correct their FHP, the classic Yang's 24 Forms of Tai Chi has been improved. The movements are mostly upper limb movements and the lower limb movements have been simplified to make the movements easy to learn. The modified Tai Chi exercise retains the traditional Tai Chi movements but is simple and easy to learn; at the same time, it increases the movement of the shoulder and neck joints. The subjects performed each exercise session in a group setting at the school gymnasium, with a professional Tai Chi instructor guiding them through a warm-up session, followed by a Tai Chi exercise session.
  Arms: Tai Chi
Behavioral: Tai Chi and Manual therapy — Intervention content of MSG included 15-min Tai Chi exercise and 15-min manual therapy, with the order of intervention being Tai Chi exercise first and then manual therapy.
  Arms: Tai Chi and Manual therapy

SUMMARY:
Forward head posture (FHP) is a prevalent deformity that can cause various health issues in adolescents. The programs combining manual therapy (MT) and stability exercises (SE) have shown better effectiveness than stability exercises and home exercises in recovering FHP. However, the effectiveness of the therapy program consisting of Tai Chi and MT for recovering FHP remains unclear. Therefore, this study aimed to investigate the effects of Tai Chi with MT on FHP recovery. Meanwhile, with a particular focus on personalized medicine, we utilized explainable artificial intelligence (XAI) to predict if individuals would reverse to healthy posture based on different interventions.

ELIGIBILITY:
Inclusion Criteria:

1. who was diagnosed as FHP;
2. whose age was between ten to nineteen years old.

Exclusion Criteria:

1. who had nervous system disease or musculoskeletal system disease;
2. who had congenital scoliosis or congenital malformation disease;
3. who participated in other sports training;
4. who participated in other training program in the past of three months before the beginning of the study.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Using photogrammetry to calculate the cranial vertebral angle of participants before and after the intervention. | Month 3
  Participants' cranial vertebral angles before and after the intervention will be measured using photogrammetry to assess the change in cranial vertebral angle at 3 months compared to baseline.
Using universal goniometer to calculate the cervical range of motion of participants before and after the intervention. | Month 3
  Participants' cervical range of motion before and after the intervention will be measured using universal goniometer to assess the change in cranial vertebral angle at 3 months compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Center of Exercise Epidemiology, Changchun, Jilin, China